CLINICAL TRIAL: NCT03738007
Title: A Randomized, Multi Center, Single-blind, Active-controlled, Matched Pairs Design Clinical Study to Evaluate the Correction of Facial Wrinkles and Folds and Safety of HA IDF II Versus Perlane in Nasolabial Fold Injection
Brief Title: Clinical Study to Evaluate the Correction of Facial Wrinkles and Folds and Safety of YVOIRE Volume Versus Perlane in Nasolabial Fold Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-HACL009
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Temporary Correction of Wrinkles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA IDF II (Experimental)
  Interventions: Device: HA IDF II
- Perlane (Active Comparator)
  Interventions: Device: Perlane

INTERVENTIONS:
Device: HA IDF II — Treatment with HA IDF II (YVOIRE volume)
  Arms: HA IDF II
Device: Perlane — Treatment with Perlane
  Arms: Perlane

SUMMARY:
This study was purposed to evaluate the non-inferiority of YVOIRE volume, a hyaluronic acid product, in terms of correction of wrinkles and safety in nasolabial fold deep-dermal injection, compared to Perlane, the control preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Women in 30~55 years.
2. Those whose wrinkle scores in the treatment site (nasolabial fold) at the screening visit were Stage 3 or 4 in the 5-stage Wrinkle Severity Rating Scale (WSRS) symmetrically
3. Those who were informed on this study in detail, understood it completely, decided to participate in the study own their own and signed on the informed consent form.

Exclusion Criteria:

1. Those with a skin disease in the face (skin infection, eczema, psoriasis, rosacea, herpes etc.)
2. Those with a history of severe allergy
3. Those with hypertrophic scar or a history of kelloid
4. Patients with an autoimmune disease
5. Those with hepatic dysfunction or abnormality in coagulation, or those administering an anticoagulant (aspirin, warfarin etc.) concomitantly
6. Those who had used a local topical preparation (steroid, retinoid) within 4 weeks prior to the study
7. Those who had underwent a chemical peeling, laser procedure (including IPL) or insertion of other bioadaptive materials (however, those who had been treated with HA filler could participate in the study if the date of treatment was known and the investigator judged that the filler effect had disappeared).
8. Patients with a malignant tumor
9. Women in pregnancy or lactation
10. Hepatitis carriers or VDRL/HIV positive patients
11. Those with a hypersensitivity to the investigational medical device of this study
12. Other persons including those considered as difficult to perform this study by the principal investigator

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Average of Wrinkle Severity Rating Scale (WSRS) score evaluated by the evaluating investigator at Week 26 (Visit 7) after the final treatment with the investigational medical device. | Week 26 (Visit 7)
  Wrinkle Severity Rating Scale (WSRS)
  1. Absent: no visible fold; continuous line
  2. Mild: Shallow but visible fold with slight indentation; minor facial feature
  3. Moderate: moderately deep fold; clear facial feature visible at normal appearance but not when stretched. Excellent correction expected.
  4. Severe: very long and deep; prominent facial feature; less than 2mm visible fold when stretched
  5. Extreme: extremely deep and long folds; 2-4mm visible v-shaped fold when stretched; detrimental to appearance; unlikely to have satisfactory correction with injectable implant alone